CLINICAL TRIAL: NCT06441370
Title: Patient Satisfaction With Physiological Childbirth in Water or on Land a Prospective Study at the Tourcoing Hospital Maternity Unit
Brief Title: Patient Satisfaction During Physiological Water or Land Birth: a Prospective Study in an French Tertiary Maternity Unit.
Acronym: AQUAMODA
Status: Recruiting | Type: Observational
Sponsor: Tourcoing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 22.01415.000084
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Water Birth
MeSH Terms: interventions — Natural Childbirth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women with water births
  Interventions: Procedure: waterbirth
- women giving birth on land

INTERVENTIONS:
Procedure: waterbirth — waterbirth: laboured for all or part of the first stage of labour and remained in the water for birth of newborn
  Groups: women with water births

SUMMARY:
A study will be carried out to compare the level of satisfaction and psychological state of women who give birth in water with those who give birth out of water.

The aim is to demonstrate the benefits of water birth and justify its place in the healthcare offering.

ELIGIBILITY:
Inclusion Criteria:

* Major patient
* Social security beneficiary
* Presence of a companion
* Delivery greater than or equal to 37 weeks of amenorhoea
* Spontaneous labor
* Cephalic presentation
* Physiological delivery by woman's choice according to 2017 HAS criteria (French recommendations)

Exclusion Criteria:

* Patient under court protection
* Patient under guardianship or curatorship
* Placement of an epidural
* Language barrier
* Unexpected delivery (unwanted by the woman)
* Scarred uterus
* Meconium fluid
* Maternal pathologies: epilepsy, MS (depending on neurological opinion), diabetes (types 1 and 2), herpes infection, HIV, HBV, HCV
* History of delivery hemorrhage > 1L
* History of shoulder dystocia/clavicle fracture
* Metrorrhagia
* Administration of nalbuphine within 2 hours of birth.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who have chosen to give birth physiologically at the Maternity unit will be offered the study during their maternity stay.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Perceived control over childbirth | This questionnaire will be achieved by participating women within 3 days postpartum, before discharge from the maternity ward.
  The "perception of control over childbirth" dimension of the QEVA (Quality and Experience of Childbirth), a long version with a total of 6 dimensions. The score associated with the "perception of control over childbirth" dimension is obtained by averaging responses to items 8, 10, 11, 12, 14 and 18 of the questionnaire. The response to each of these items is coded on a Likert scale from 1 to 4, with a high value corresponding to poor control.

SECONDARY OUTCOMES:
Dimension of the quality and experience of childbirth within 3 days of delivery | This questionnaire is to be completed within 3 days of delivery, before discharge from the maternity hospital.
  The scores associated with the 5 other dimensions of the QEVA questionnaire:
  * Expectations, defined by items 9, 15 and 20;
  * Sensory experience, defined by items 3 and 16;
  * Relationship with caregivers, defined by items 5, 6, 7 and 13;
  * Emotions, defined by items 1, 2, 4, 21, 22, 23 and 24;
  * First moments with baby, defined by items 17, 18 and 19; Answers to the questions are coded on Likert scales from 1 to 4. Each score is calculated by averaging the responses to the questions in the dimension in question.
Dimension of the quality and experience of childbirth within 2 months of delivery | This questionnaire is to be completed within 2 months of delivery.
  The scores associated with the 5 other dimensions of the QEVA questionnaire:
  * Expectations, defined by items 9, 15 and 20;
  * Sensory experience, defined by items 3 and 16;
  * Relationship with caregivers, defined by items 5, 6, 7 and 13;
  * Emotions, defined by items 1, 2, 4, 21, 22, 23 and 24;
  * First moments with baby, defined by items 17, 18 and 19; Answers to the questions are coded on Likert scales from 1 to 4. Each score is calculated by averaging the responses to the questions in the dimension in question.
Anxiety and depression at 2 months of delivery. | This questionnaire is to be completed within 2 months of delivery.
  The Edinburgh Postnatal Depression Scale (EPDS) will be used to assess anxiety and depression and depression at 2 months postpartum in order to screen for possible postpartum depression.

CONTACTS AND LOCATIONS:
Overall Officials: GOBERT JG julia, MD, Principal Investigator — Tourcoing Hospital; GAILLARD JG Julie, Principal Investigator — Tourcoing Hospital
Locations (1):
- Tourcoing Hospital, Tourcoing, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No